CLINICAL TRIAL: NCT04990804
Title: Opioid Free vs. Standard Perioperative Pain Regimen for Anterior Cervical Discectomy and Fusion (ACDF) Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Limitations of the prospective study design revealed that a retrospective study design would be better suited.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Cervical Spine Research Society (Other)
Responsible Party: Principal Investigator, Amir Abtahi, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210432
Record Dates: First submitted 2021-07-29; First posted 2021-08-05 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use; Spinal Diseases; Surgery--Complications; Surgery; Postoperative Pain
MeSH Terms: conditions — Spinal Diseases; Pain, Postoperative | interventions — Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: Randomized, Non-Blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Perioperative Pain Regimen (Active Comparator): Patients will be provided a prescription for low dose opioids for 5 days postoperatively (Hydrocodone/Acetaminophen 5/325mg or Oxycodone/Acetaminophen 5/325mg) to be taken every 6 hours as needed for pain. Refills may be provided (Hydrocodone/Acetaminophen 5/325mg or Oxycodone/Acetaminophen 5/325mg) if requested by the patient at the providers discretion. In addition, patients will also be prescribed Gabapentin 300mg q8 hours or Pregabalin 75mg twice daily and a muscle relaxer (Methocarbamol 750mg BID or Flexeril 5-10 mg TID) as needed for spasms. Alternative muscle relaxers (Metaxalone 800 mg TID or Tizanidine 2-6 mg TID) may be utilized if contraindications to methocarbamol and cyclobenzaprine exist.
  Interventions: Drug: Opioid Analgesic
- Opioid-Free Perioperative Pain Regimen (Experimental): Patients will receive no opioids. Pain will be managed with Acetaminophen 1000mg q8 hours, Ketorolac 10mg every 6 hours (for 5 days), Gabapentin 300mg q8 hours or Pregabalin 75mg twice daily, and a muscle relaxer (Methocarbamol 750mg BID or Cyclobenzaprine 5-10 mg TID) all to be taken as scheduled for the first 2 weeks (except Ketorolac - 5 days) postoperatively as side effects permit. Other NSAIDS (Naprosyn 500 mg BID or Ibuprofen 800 mg TID) may be utilized if contraindications to Ketorolac exist. Famotidine (20mg BID) or Omeprazole (20mg daily) will be prescribed along with NSAIDS for GI prophylaxis. Alternative muscle relaxers (Metaxalone 800 mg TID or Tizanidine 2-6 mg TID) may be utilized if contraindications to methocarbamol and cyclobenzaprine exist.
  Interventions: Drug: Opioid-Free Postoperative Pain Regimen

INTERVENTIONS:
Drug: Opioid Analgesic — Patients will be provided a prescription for low dose opioids for 5 days postoperatively (Hydrocodone/Acetaminophen 5/325mg or Oxycodone/Acetaminophen 5/325mg) to be taken every 6 hours as needed for pain. Refills may be provided (Hydrocodone/Acetaminophen 5/325mg or Oxycodone/Acetaminophen 5/325mg) if requested by the patient at the providers discretion. In addition, patients will also be prescribed Gabapentin 300mg q8 hours or Pregabalin 75mg twice daily and a muscle relaxer (Methocarbamol 750mg BID or Flexeril 5-10 mg TID) as needed for spasms. Alternative muscle relaxers (Metaxalone 800 mg TID or Tizanidine 2-6 mg TID) may be utilized if contraindications to methocarbamol and cyclobenzaprine exist.
  Arms: Standard Perioperative Pain Regimen
Drug: Opioid-Free Postoperative Pain Regimen — Patients will receive no opioids. Pain will be managed with Acetaminophen 1000mg q8 hours, Ketorolac 10mg every 6 hours (for 5 days), Gabapentin 300mg q8 hours or Pregabalin 75mg twice daily, and a muscle relaxer (Methocarbamol 750mg BID or Cyclobenzaprine 5-10 mg TID) all to be taken as scheduled for the first 2 weeks (except Ketorolac - 5 days) postoperatively as side effects permit. Other NSAIDS (Naprosyn 500 mg BID or Ibuprofen 800 mg TID) may be utilized if contraindications to Ketorolac exist. Famotidine (20mg BID) or Omeprazole (20mg daily) will be prescribed along with NSAIDS for GI prophylaxis. Alternative muscle relaxers (Metaxalone 800 mg TID or Tizanidine 2-6 mg TID) may be utilized if contraindications to methocarbamol and cyclobenzaprine exist.
  Arms: Opioid-Free Perioperative Pain Regimen

SUMMARY:
Patients undergoing 1-3 level Anterior Cervical Discectomy and Fusion (ACDF) at the levels between C2 and T1 will be enrolled into this randomized prospective study. All patients enrolled in this study will undergo a trial of non-surgical treatment prior to the recommendation for surgery. After enrollment, patients will be randomized utilizing a block randomization strategy to one of two treatment groups - a standard opioid-containing postoperative pain regimen versus a non-opioid postoperative pain regimen. Postoperative outcomes will be assessed.

DETAILED DESCRIPTION:
Patients will be followed for 12 months and the following Specific Aims will be assessed:

Aim 1: Evaluate whether utilization of a non-opioid postoperative pain regimen after ACDF leads to lower rates of new chronic opioid use when compared with postoperative pain regimens utilizing opioids.

Aim 2: Evaluate whether utilization of a non-opioid postoperative pain regimen after ACDF results in equivalent postoperative pain scores in the early postoperative period.

Aim 3: Evaluate whether utilization of a non-opioid postoperative pain regimen after ACDF leads to equivalent clinical outcomes when compared with postoperative pain regimens utilizing opioids at 3 months and 12 months.

Aim 4: Evaluate whether utilization of a non-opioid postoperative pain regimen after ACDF leads to fewer postoperative complications when compared with postoperative pain regimens utilizing opioids.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of degenerative cervical spine disease
* Failure of conservative therapy
* Age ≥18 years
* Skeletal maturity.

Exclusion Criteria:

* Preoperative chronic opioid use as determined by self report (>45 out of past 90 days)
* History of chronic kidney disease
* Revision cervical spine surgery
* Concurrent posterior cervical fusion
* Does the patient have an intolerance to NSAIDs (non-steroidal anti-inflammatory drugs)?
* Does the patient have any preexisting health condition the study physician believes will be exacerbated by participating in this study?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Perioperative Pain Regimen | Opioid-Free Perioperative Pain Regimen
Started | 5 | 3
Completed | 4 | 2
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Perioperative Pain Regimen | Opioid-Free Perioperative Pain Regimen | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: New Chronic Opioid Use
Description: Opioid prescription for > or = 45 days in 90 day window (9-12 months postoperatively)
Time Frame: 9-12 months
Population: There is no data to analyze for this outcome, as patients were not contacted at the specified time point and no data was collected. Data was not collected due to early termination of the study.
Arm/Group | Standard Perioperative Pain Regimen | Opioid-Free Perioperative Pain Regimen
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Postoperative Pain
Description: Numeric Rating Scale (NRS) arm pain and neck pain scores. This scale grades pain on a scale from 0 to 10, with 0 being no pain and 10 being the worst pain imaginable. The higher the pain score, the more ineffective a patient's pain medication regimen is.
Time Frame: Postoperative day 1, 7, 14
Population: One participant in the Standard Perioperative Pain Regimen group was lost to follow-up after randomization. One participant in the Opioid-Free Perioperative Pain Regimen group was lost to follow-up after randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Perioperative Pain Regimen | Opioid-Free Perioperative Pain Regimen
Number analyzed (Participants) | 4 | 2
score on a scale
  Current Neck Pain Day 1 | 4.0 (2.9) | 1.5 (0.7)
  Current Neck Pain Day 7 | 4.2 (2.4) | 0.0 (0.0)
  Current Neck Pain Day 14: number analyzed (Participants) | 4 | 1
  Current Neck Pain Day 14 | 2.0 (3.4) | 4.0
  Average Neck Pain Day 1 | 5.5 (4.1) | 1.5 (0.7)
  Average Neck Pain Day 7 | 5.3 (3.6) | 0.0 (0.0)
  Average Neck Pain Day 14 | 3.8 (3.3) | 1.5 (2.1)
  Current Arm Pain Day 1 | 2.5 (5.0) | 0.5 (0.7)
  Current Arm Pain Day 7 | 1.8 (3.5) | 1.5 (0.7)
  Current Arm Pain Day 14 | 1.8 (3.5) | 3.0 (1.4)
  Average Arm Pain Day 1 | 0.5 (0.7) | 3.0 (4.8)
  Average Arm Pain Day 7 | 1.0 (0.0) | 1.8 (3.5)
  Average Arm Pain Day 14 | 2.5 (0.7) | 2.0 (4.0)

3. Secondary Outcome: PROMIS-29 (Patient-Reported Outcomes Measurement Information System)
Description: A disease non-specific tool for measuring medication management, depression, anxiety, fatigue, pain interference, sleep disturbance, and phsyical functioning. Each domain contains questions specific to what trait is being measure. Scores have a mean of 50 and a standard deviation of 10. The higher the score, the better the outcome.
Time Frame: 3 and 12 months postoperatively
Population: as for outcome 1
Arm/Group | Standard Perioperative Pain Regimen | Opioid-Free Perioperative Pain Regimen
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Neck Disability Index (NDI)
Time Frame: 3 and 12 months postoperatively
Population: as for outcome 1
Arm/Group | Standard Perioperative Pain Regimen | Opioid-Free Perioperative Pain Regimen
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Return to Work Status
Time Frame: 3 and 12 months postoperatively
Population: as for outcome 1
Arm/Group | Standard Perioperative Pain Regimen | Opioid-Free Perioperative Pain Regimen
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient Satisfaction With the Surgical Outcome
Description: Ask the patient how satisfied they are will their surgical treatment and includes the following responses. 1. Very satisfied 2. Somewhat satisfied 3. Neither satisfied nor dissatisfied 4. Somewhat dissatisfied 5. Very dissatisfied
Time Frame: 3 and 12 months postoperatively
Population: as for outcome 1
Arm/Group | Standard Perioperative Pain Regimen | Opioid-Free Perioperative Pain Regimen
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Postoperative Adverse Events
Description: Readmissions, adverse events, serious adverse events
Time Frame: Baseline to 12 months
Population: as for outcome 1
Arm/Group | Standard Perioperative Pain Regimen | Opioid-Free Perioperative Pain Regimen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to study termination - approximately 6 months
Arm/Group | Standard Perioperative Pain Regimen | Opioid-Free Perioperative Pain Regimen
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT04990804/Prot_SAP_000.pdf